CLINICAL TRIAL: NCT06366126
Title: Long Term Impact of Child Abuse in University Students
Status: Completed | Type: Observational
Sponsor: Delta University for Science and Technology (Other)
Responsible Party: Principal Investigator, Amira Hussin Hussin Mohammed, Assistant professor at faculty of physical therapy, Delta University for Science and Technology
Other Study IDs: Child Abuse
Record Dates: First submitted 2024-04-10; First posted 2024-04-15 (Actual); Last update posted 2024-04-15 (Actual); Status verified 2024-04

CONDITIONS: Child Abuse

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Based on research and studies, a broad conceptualization of child abuse and neglect has progressively been constructed, defining it as all actions carried out by caregivers that significantly interfere in the child's optimum development and do not adhere to social standards. This conceptualization contemplates aspects such as neglecting physical-biological, cognitive, emotional, and social needs, and the different types of child maltreatment are also classified.

This study aimed too evaluate the psychological and social long-term effects of different types of child abuse.

ELIGIBILITY:
* Inclusion criteria:

  1. University students passed through the experience of being abused in their childhood
  2. Males and females
  3. Residing in urban or rural area in Al Dakahleya governorate- Egypt
* Exclusion criteria:

  * Individuals with no or questionable history of child abuse

Ages: 18 Years to 23 Years | Sex: All
Age Groups: Adult
Study Population: A random sample of 242 participants from university students with history of exposure to child abuse in Al Dakahleya governorate, Egypt, consisted of 151 Males and 91 Females
Sampling Method: Probability Sample
Enrollment: 242 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
tailored questionnaire | At the baseline of evaluation
  type and physical, social and psycho behavioral long term impact of child abuse

CONTACTS AND LOCATIONS:
Locations (1):
- Amira Hussin Mohammed, Gamasa, Egypt

IPD SHARING:
Plan to Share IPD: No